CLINICAL TRIAL: NCT01316614
Title: Randomized Controlled Trial of Endoscopic Ultrasound Guided Fine Needle Aspiration of Solid Lesions With and Without a Stylet
Brief Title: EUS-guided Fine Needle Aspiration (FNA) With and Without the Use of a Stylet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201105404
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Biopsy, Fine-Needle; Biopsy, Fine-Needle/Methods; Endosonography
Keywords: Fine-Needle Aspiration; Stylet; Solid Mass; Endoscopic Ultrasound (EUS)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- With Stylet & Without Stylet (Experimental): There will only be one arm in this study. This arm will undergo EUS-guided FNA with the use of a stylet for half of their FNA passes and without a stylet for the other half. Patients will be exposed to an equal number of passes with and without a stylet. Each pass will be individually assessed by a skilled cytopathologist who is blinded to the technique used. We will compare the adequacy of both techniques to determine whether or not a stylet leads to a higher diagnostic accuracy rate in patients with solid lesions.
  Interventions: Device: FNA with and without a stylet

INTERVENTIONS:
Device: FNA with and without a stylet — If the patient agrees to enrollment in the study, the initial stage of the EUS exam will be performed in the usual manner. If a solid lesion that requires FNA is identified, an envelope will be opened which contains a computer generated randomization sequence for all passes. These sequences will be generated by a web-based program at http://www.randomizer.org/form.htm. Passes will be made based on the randomization, either with or without a stylet. Six passes (three with a stylet and three without a stylet) will be performed on solid lesions and four passes (two with and two without a stylet) will be performed on lymph nodes. Additional passes will be made at the discretion of the endosonographer as clinically indicated but will not be included in the data.
  Other Names: Cook Medical EchoTip® Ultra Endoscopic Ultrasound Needles

SUMMARY:
The purpose of this study is to determine that there is no difference in final diagnosis of FNA specimens without a stylet, compared to using a stylet, when examined by a skilled cytopathologist.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS)-guided fine needle aspiration (FNA) is a highly accurate method for cytologic diagnosis of malignancy and is routinely performed to diagnose and stage pancreatobiliary, esophageal, gastric, rectal malignancies and subepithelial gastrointestinal lesions. There are variations in EUS-FNA technique including the use of suction, the area of the lesion to target (center versus periphery), gauge of needle, and use of a stylet.

The stylet is a metal wire which is included in the needle assembly. The use of a stylet is used purely for mechanical purposes, not for the protection or safety of the patients. It is thought that the stylet prevents the needle from becoming clogged with gastrointestinal epithelial cells or mucus. To our knowledge, comparing the diagnostic accuracy of EUS-FNA with a stylet to the accuracy without a stylet has not been studied.

The optimal technique for EUS-FNA has not been established. The reported accuracy rate of EUS-FNA (which contains heterogeneous sampling techniques, including with and without a stylet) is 71-98% for pancreatic masses, 90% for lymph nodes, and 67-92% for submucosal gastrointestinal lesions. Typically, FNA is performed with or without a stylet using a 22 gauge or 25 gauge needle with similar diagnostic accuracy.

When the target lesion is identified, the needle is advanced through the gastrointestinal wall into the lesion under ultrasound guidance. If a stylet is being used, it is removed at this point. A 10 cc syringe under suction is then placed on the end of the needle assembly and the needle is moved back and forth within the lesion to gather cells. The assembly is then removed and the needle contents are expelled onto slides and into preservative media. The stylet is then reinserted and the needle assembly is advanced through the scope for another pass. In the absence of on-site cytopathology, 7 passes with or without a stylet of a solid lesion and 5 passes of lymph nodes with or without a stylet are recommended to achieve high diagnostic accuracy.

EUS-FNA is time consuming, mainly because the stylet needs to be carefully reinserted through the needle prior to each pass. Theoretically, the use of a stylet prevents clogging of the needle with gastrointestinal epithelial cells and mucus which can affect the adequacy of the specimen. However, there are no data to support this. As such there is a variation in practice patterns, with some endosonographers who routinely use a stylet and those that do not. Additionally, those who perform percutaneous FNA frequently do so using needles that do not have a stylet. A recent study suggests that the use of a stylet improves diagnostic accuracy in percutaneous FNA of thyroid lesions. To our knowledge, there have been no studies assessing the use of a stylet on tissue adequacy in EUS-guided FNA.

If the practice of using a stylet during EUS-guided FNA is found to yield the same number of adequate tissue samples as those done without a stylet, then the use of a stylet would be an unnecessary. As stylet replacement is the most time consuming step in FNA, the time of the procedure could be shortened significantly if the stylet is not required.

We propose a randomized controlled trial of EUS guided FNA with and without stylet which will help determine whether the use of a stylet is integral in obtaining adequate tissue aspirates in the diagnosis of solid lesions. To our knowledge, there have been no prospective, randomized studies addressing the effect of the presence or absence of a stylet on specimen adequacy during EUS-guided FNA.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the Washington University Interventional Endoscopy Division for EUS-guided FNA of a solid lesion (e.g. pancreatic mass, gastric wall mass, or lymphadenopathy)

Exclusion Criteria:

* Patients <18 years of age
* patients who cannot provide independent informed consent (i.e. patients with dementia or with a health care proxy)
* pregnant women (as determined by pregnancy test given as part of standard of care)
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Mullady, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Wiersema MJ, Vilmann P, Giovannini M, Chang KJ, Wiersema LM. Endosonography-guided fine-needle aspiration biopsy: diagnostic accuracy and complication assessment. Gastroenterology. 1997 Apr;112(4):1087-95. doi: 10.1016/s0016-5085(97)70164-1. PMID 9097990
- [Background] Harewood GC, Wiersema MJ. Endosonography-guided fine needle aspiration biopsy in the evaluation of pancreatic masses. Am J Gastroenterol. 2002 Jun;97(6):1386-91. doi: 10.1111/j.1572-0241.2002.05777.x. PMID 12094855
- [Background] Chhieng DC, Jhala D, Jhala N, Eltoum I, Chen VK, Vickers S, Heslin MJ, Wilcox CM, Eloubeidi MA. Endoscopic ultrasound-guided fine-needle aspiration biopsy: a study of 103 cases. Cancer. 2002 Aug 25;96(4):232-9. doi: 10.1002/cncr.10714. PMID 12209665
- [Background] Eloubeidi MA, Chen VK, Eltoum IA, Jhala D, Chhieng DC, Jhala N, Vickers SM, Wilcox CM. Endoscopic ultrasound-guided fine needle aspiration biopsy of patients with suspected pancreatic cancer: diagnostic accuracy and acute and 30-day complications. Am J Gastroenterol. 2003 Dec;98(12):2663-8. doi: 10.1111/j.1572-0241.2003.08666.x. PMID 14687813
- [Background] Savides TJ, Donohue M, Hunt G, Al-Haddad M, Aslanian H, Ben-Menachem T, Chen VK, Coyle W, Deutsch J, DeWitt J, Dhawan M, Eckardt A, Eloubeidi M, Esker A, Gordon SR, Gress F, Ikenberry S, Joyce AM, Klapman J, Lo S, Maluf-Filho F, Nickl N, Singh V, Wills J, Behling C. EUS-guided FNA diagnostic yield of malignancy in solid pancreatic masses: a benchmark for quality performance measurement. Gastrointest Endosc. 2007 Aug;66(2):277-82. doi: 10.1016/j.gie.2007.01.017. PMID 17643700
- [Background] Eloubeidi MA, Jhala D, Chhieng DC, Chen VK, Eltoum I, Vickers S, Mel Wilcox C, Jhala N. Yield of endoscopic ultrasound-guided fine-needle aspiration biopsy in patients with suspected pancreatic carcinoma. Cancer. 2003 Oct 25;99(5):285-92. doi: 10.1002/cncr.11643. PMID 14579295
- [Background] Vander Noot MR 3rd, Eloubeidi MA, Chen VK, Eltoum I, Jhala D, Jhala N, Syed S, Chhieng DC. Diagnosis of gastrointestinal tract lesions by endoscopic ultrasound-guided fine-needle aspiration biopsy. Cancer. 2004 Jun 25;102(3):157-63. doi: 10.1002/cncr.20360. PMID 15211474
- [Background] Mitsuhashi T, Ghafari S, Chang CY, Gu M. Endoscopic ultrasound-guided fine needle aspiration of the pancreas: cytomorphological evaluation with emphasis on adequacy assessment, diagnostic criteria and contamination from the gastrointestinal tract. Cytopathology. 2006 Feb;17(1):34-41. doi: 10.1111/j.1365-2303.2006.00277.x. PMID 16417563
- [Background] Siddiqui UD, Rossi F, Rosenthal LS, Padda MS, Murali-Dharan V, Aslanian HR. EUS-guided FNA of solid pancreatic masses: a prospective, randomized trial comparing 22-gauge and 25-gauge needles. Gastrointest Endosc. 2009 Dec;70(6):1093-7. doi: 10.1016/j.gie.2009.05.037. Epub 2009 Jul 28. PMID 19640524
- [Background] LeBlanc JK, Ciaccia D, Al-Assi MT, McGrath K, Imperiale T, Tao LC, Vallery S, DeWitt J, Sherman S, Collins E. Optimal number of EUS-guided fine needle passes needed to obtain a correct diagnosis. Gastrointest Endosc. 2004 Apr;59(4):475-81. doi: 10.1016/s0016-5107(03)02863-3. PMID 15044881
- [Background] Cappelli C, Pirola I, Gandossi E, De Martino E, Agosti B, Castellano M. Fine-needle aspiration cytology of thyroid nodule: does the needle matter? South Med J. 2009 May;102(5):498-501. doi: 10.1097/SMJ.0b013e31819c7343. PMID 19373168
- [Background] Erickson RA, Sayage-Rabie L, Beissner RS. Factors predicting the number of EUS-guided fine-needle passes for diagnosis of pancreatic malignancies. Gastrointest Endosc. 2000 Feb;51(2):184-90. doi: 10.1016/s0016-5107(00)70416-0. PMID 10650262
- [Background] Gonen M. Sample size and power for McNemar's test with clustered data. Stat Med. 2004 Jul 30;23(14):2283-94. doi: 10.1002/sim.1768. PMID 15236431
- [Background] Obuchowski NA. On the comparison of correlated proportions for clustered data. Stat Med. 1998 Jul 15;17(13):1495-507. doi: 10.1002/(sici)1097-0258(19980715)17:133.0.co;2-i. PMID 9695194
- [Background] Nguyen YP, Maple JT, Zhang Q, Ylagan LR, Zhai J, Kohlmeier C, Jonnalagadda S, Early DS, Edmundowicz SA, Azar RR. Reliability of gross visual assessment of specimen adequacy during EUS-guided FNA of pancreatic masses. Gastrointest Endosc. 2009 Jun;69(7):1264-70. doi: 10.1016/j.gie.2008.08.030. Epub 2009 Feb 24. PMID 19243768
- [Derived] Wani S, Early D, Kunkel J, Leathersich A, Hovis CE, Hollander TG, Kohlmeier C, Zelenka C, Azar R, Edmundowicz S, Collins B, Liu J, Hall M, Mullady D. Diagnostic yield of malignancy during EUS-guided FNA of solid lesions with and without a stylet: a prospective, single blind, randomized, controlled trial. Gastrointest Endosc. 2012 Aug;76(2):328-35. doi: 10.1016/j.gie.2012.03.1395. Epub 2012 Jun 12. PMID 22695205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 07/21/2010 and closed to participant enrollment on 02/07/2012.
Groups:
- With Stylet & Without Stylet: There will only be one arm in this study. This arm will undergo EUS-guided FNA with the use of a stylet for half of their FNA passes and without a stylet for the other half. Patients will be exposed to an equal number of passes with and without a stylet. Only the order of the passes were randomized.
Period: Overall Study
Arm/Group | With Stylet & Without Stylet
Started | 137
Completed | 100
Not Completed | 37
Not completed — No solid lesion and FNA not indicated | 25
Not completed — Cytology slides not available for review | 4
Not completed — Cystic lesion | 5
Not completed — Inadequate number of passes | 2
Not completed — Medically unstable | 1

BASELINE CHARACTERISTICS:
Groups:
- With Stylet & Without Stylet: There will only be one arm in this study. This arm will undergo EUS-guided FNA with the use of a stylet for half of their FNA passes and without a stylet for the other half. Patients will be exposed to an equal number of passes with and without a stylet.
Arm/Group | With Stylet & Without Stylet
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 87
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Lesions that underwent EUS-FNA [Number; unit: participants]
  Pancreatic masses | 58
  Lymph nodes | 25
  Gastric subepithelial lesion | 6
  Esophageal subepithelial lesion | 2
  Biliary stricture | 3
  Hilar mass | 1
  Liver | 1
  Ampulla | 1
  Left adrenal gland | 1
  Mediastinal mass | 2
Size of lesions [Mean (Standard Deviation); unit: centimeters (cm)]
  All lesions | 2.95 (21.8)
  Pancreas | 3.18 (1.53)
  Lymph node | 2.08 (1.3)
  All other lesions | 3.35 (4.0)
Tissue echogenecity [Number; unit: participants]
  Hypoechoic | 86
  Mixed echogenicity | 14
Needle gauge used [Number; unit: participants]
  22-gauge | 77
  25-gauge | 23

OUTCOME MEASURES:

1. Primary Outcome: Compare Adequacy of Diagnoses in Passes With and Without a Stylet
Description: The number of passes was determined by the lesion site and mirrored clinical practice (6 passes for pancreatic/other lesions and 4 passes for lymph nodes). The order of these passes was determined by a preprinted randomization sequence kept in an opaque sealed envelope that was opened by the research coordinator or EUS technologist after enrollment. Each participant had an equal number of passes with stylet and without stylet.
  There was no communication between the endosonographer and the cytopathologist regarding the adequacy of the specimen or diagnosis until all passes had been completed. The on-site evaluation of smears was performed to assess cellular adequacy and to assess the need for any additional passes. Additional passes were made at the discretion of the endosonographer as clinically indicated but were not included in the final analysis. The cytology slides were evaluated by 3 experienced cytopathologists who were all blinded to the stylet status of the passes.
Time Frame: At the time of EUS-FNA procedure (Day 1)
Population: 100 participants were analyzed. Each participant had an equal number of passes with a stylet and without a stylet. 275 overall passes were performed with a stylet and 275 passes were performed without a stylet. The actual passes are represented in the table.
Measure: Number; unit: passes
Groups:
- With Stylet: Each participant had half of their passes performed with a stylet.
- Without Stylet: Each participant had half of their passes performed without a stylet.
Arm/Group | With Stylet | Without Stylet
Number analyzed (Participants) | 100 | 100
passes
  Benign or negative for malignancy | 80 | 68
  Atypical | 21 | 18
  Suspicious | 23 | 15
  Malignant | 94 | 110
  Inadequate for reporting | 57 | 64

2. Secondary Outcome: Degree of Cellularity
Description: Percentage of area of slide that contains cells of the representative lesion
Time Frame: At the time of EUS-FNA procedure (Day 1)
Population: 100 participants were analyzed. Each participant had an equal number of passes with a stylet and without a stylet. 275 passes were performed with a stylet and 275 passes were performed without a stylet. The actual passes are represented in the table.
Measure: Number; unit: passes
Arm/Group | With Stylet | Without Stylet
Number analyzed (Participants) | 100 | 100
passes
  No representative cells present | 66 | 72
  Representative cells present in <25% | 58 | 46
  Representative cells present in <25-50% slide | 97 | 99
  Representative cells present in >50% of the slide | 54 | 58

3. Secondary Outcome: Degree of Cellularity
Description: Number of cells per slide
Time Frame: At the time of EUS-FNA procedure (Day 1)
Population: as for outcome 2
Measure: Number; unit: passes
Arm/Group | With Stylet | Without Stylet
Number analyzed (Participants) | 100 | 100
passes
  Fair (<100 cells/slide) | 127 | 120
  Good (100-1000 cells/slide) | 70 | 82
  Excellent (>1000 cells/slide) | 78 | 73

4. Secondary Outcome: Adequacy of Specimen
Time Frame: At the time of EUS-FNA procedure (Day 1)
Population: as for outcome 2
Measure: Number; unit: passes
Arm/Group | With Stylet | Without Stylet
Number analyzed (Participants) | 100 | 100
passes
  Inadequate | 87 | 78
  Adequate | 188 | 197

5. Secondary Outcome: Contamination
Description: Percentage of area of slide that represents GI contamination
Time Frame: At the time of EUS-FNA procedure (Day 1)
Population: as for outcome 2
Measure: Number; unit: passes
Arm/Group | With Stylet | Without Stylet
Number analyzed (Participants) | 100 | 100
passes
  No contaminations seen | 212 | 220
  Contamination present in <25% of the slide | 52 | 47
  Contamination present in 25%-50% of the slide | 7 | 5
  Contamination present in >50% of the slide | 4 | 3

6. Secondary Outcome: Amount of Blood
Time Frame: At the time of EUS-FNA procedure (Day 1)
Population: as for outcome 2
Measure: Number; unit: passes
Arm/Group | With Stylet | Without Stylet
Number analyzed (Participants) | 100 | 100
passes
  Minimal | 126 | 120
  Moderate | 82 | 86
  Significant | 67 | 69

ADVERSE EVENTS:
Arm/Group | With Stylet & Without Stylet
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes